CLINICAL TRIAL: NCT03971487
Title: Ocrelizumab for Psychoses Possibly Caused by Synaptic Autoimmunity
Brief Title: Ocrelizumab for Psychosis by Autoimmunity
Acronym: OPA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00021901
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Schizo-Affective Type of Psychosis; Schizophrenia
Keywords: schizo-affective psychosis; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Restraint, Physical; Electrocardiography

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled therapeutic trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ocrelizumab (Active Comparator): Two doses of 300 mg of ocrelizumab will be administered as an intravenous infusion two weeks apart.
  Interventions: Behavioral: Psychosis and cognitive assessments; Behavioral: Physical and neuro-cognitive evaluations; Diagnostic Test: Safety labs and electrocardiogram; Biological: Ocrelizumab infusion
- Placebo (Placebo Comparator): Two placebo intravenous infusions will be administered two weeks apart.
  Interventions: Behavioral: Psychosis and cognitive assessments; Behavioral: Physical and neuro-cognitive evaluations; Diagnostic Test: Safety labs and electrocardiogram

INTERVENTIONS:
Behavioral: Psychosis and cognitive assessments — Administration of MINI, PANSS and Quality of Living scales
Behavioral: Physical and neuro-cognitive evaluations — Physical, neurological and cognitive evaluations.
Diagnostic Test: Safety labs and electrocardiogram — Metabolic panel, CBC and differential, urinalysis, ECG, recreational drugs. CD19+ B-cell count.
Biological: Ocrelizumab infusion — Two IV infusions of 300 mg of ocrelizumab 2 weeks apart
  Arms: Ocrelizumab

SUMMARY:
Some people who have what doctors currently call schizophrenia or bipolar disease may actually have a brain disease caused by auto-antibodies. Auto-antibodies are produced when the normal defense mechanism of the body goes wrong and begins to attack the body, similar to "friendly fire." Auto-antibodies attack brain receptors and then the person who has this problem begins to have hallucinations and other manifestations of schizophrenia, like feeling that people can see what they are thinking and also feeling that other people do not like them. If this disease is caused by auto-antibodies, typically the person is well until they are 15 years of age or older, but seldom older than 35 years. Then, in a matter of a few months they begin to have hallucinations and the other symptoms. Doctors still do not know whether some people with schizophrenia or bipolar disease have auto-antibodies attacking their brain. For this reason, in this study some of these patients will receive a treatment that suppresses the auto-antibodies and their symptoms after treatment will be compared with the symptoms of a group of similar patients who are given a preparation that looks like the real treatment, but it is not.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either sex, 18-35 years of age.
* Having an active psychotic disorder meeting DSM-5 criteria, including a duration of at least six months, for Schizophrenia Spectrum Disorder, as defined by the Mini International Neuropsychiatric Interview (MINI).
* A total PANSS ≥ 60 and a score ≥ 4 on at least 2 of the PANSS positive symptoms.
* Normal academic performance at least until the age of 15 years and absence of psychiatric symptoms before the same age.
* Ability to assent or consent to the performance of the study and participate in testing procedures.

Exclusion Criteria:

* The dose of antipsychotic medication (if they are on one) has been changed less than two weeks prior to baseline PANSS testing (Visit 2, see below).
* Patient treated with a medication designed to suppress the immune system, other than standard analgesics or antipyretics, in the six months prior to randomization.
* Vaccinated with a live-attenuated vaccine less than 4 weeks before ocrelizumab infusion or with a non-live vaccine less than 2 weeks before infusion.
* Active infection, or history of or known presence of recurrent or chronic infection (for example, hepatitis B or C, Human Immunodeficiency Virus, syphilis, tuberculosis, PML).
* History of brain tumor, stroke, severe head trauma or multiple sclerosis.
* Active cancer, metabolic encephalopathy, severe cardiovascular or renal disease.
* In the judgment of the PI, psychosis related to substance abuse or metabolic disorders.
* Pregnancy or lactation.
* Requirement for chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
* History of or currently active primary or secondary immunodeficiency.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Contraindications to or intolerance of oral or IV corticosteroids.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Score on the Positive and Negative Syndrome Scale (PANSS) | Six months
  It measures symptoms of psychosis

SECONDARY OUTCOMES:
Score on quality of life scales for psychiatric patients | Six months
  (modified to include input by caregivers)
Score on NIH Cognitive Toolbox | Six months
  Tablet-implemented tool testing cognitive abilities, including working memory
Antipsychotic-equivalent medication ordered by patient's psychiatrist | Six months
  Dose of medications for psychosis transformed to a standard equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Masdeu, MD, PhD, Principal Investigator — HOUSTON METHODIST NEUROLOGICAL INSTITUTE
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
It is possible that anonymized data could be shared with other researchers at the conclusion of the study.

REFERENCES:
- [Background] Masdeu JC, Dalmau J, Berman KF. NMDA Receptor Internalization by Autoantibodies: A Reversible Mechanism Underlying Psychosis? Trends Neurosci. 2016 May;39(5):300-310. doi: 10.1016/j.tins.2016.02.006. Epub 2016 Apr 26. PMID 27130657
- [Background] Masdeu JC. Detecting synaptic autoantibodies in psychoses: need for more sensitive methods. Curr Opin Neurol. 2017 Jun;30(3):317-326. doi: 10.1097/WCO.0000000000000447. PMID 28234799